CLINICAL TRIAL: NCT02885311
Title: Collaborative Care for Alcohol Use Disorders in the Patient-centered Medical Home
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 15-0743; R34AA024589 (NIH)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Alcohol-Related Disorders; Alcohol Drinking; Alcoholism; Alcohol Abuse; Alcohol Use Disorders
Keywords: Drinking; Excessive drinking; Alcohol use disorders; Primary Care
MeSH Terms: conditions — Alcohol-Related Disorders; Alcohol Drinking; Alcoholism | interventions — Naltrexone; Crisis Intervention; Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- At-Risk Drinkers (AR) (Other): AR will receive feedback about their drinking and brief advice along with follow up assessments.
  Interventions: Behavioral: Brief Advice
- Problem Drinkers (PD) (Other): PD will be offered a choice of either an evidence-based behavioral intervention(Motivational Enhancement Therapy) or medication (Naltrexone) plus medication management. These participants will also receive follow up assessments.
  Interventions: Behavioral: Motivation Enhancement Therapy; Drug: Naltrexone; Behavioral: Brief Advice
- AD with physiological withdrawal (AD-W) (Other): AD-W will referred to outpatient detoxification as part of standard care, unless medically contraindicated, and will be offered medication (naltrexone) plus medication management as or an evidence-based behavioral intervention (Modified Behavioral Self-Control Therapy [MBSCT]) adapted from our two prior protocols. These participants will also receive follow up assessments.
  Interventions: Behavioral: Modified Behavioral Self-Control Therapy; Drug: Naltrexone; Behavioral: Brief Advice
- AD with complex presentation (AD-CMPLX) (Other): AD-CMPLX will receive a referral to specialty substance use disorder treatment and also receive follow up assessments.
  Interventions: Behavioral: Brief Advice; Other: Referral to specialty substance use disorder treatment

INTERVENTIONS:
Behavioral: Motivation Enhancement Therapy — Motivation Enhancement Therapy (MET) similarly allows for goal choice in treatment, and has been shown to be effective in treating a broad spectrum of drinking problems in both abstinent and non-abstinent goal conditions. The unique goals of MET (enhancing intrinsic motivation for change and facilitating development of a self-generated change plan).
  Other Names: MET
  Arms: Problem Drinkers (PD)
Behavioral: Modified Behavioral Self-Control Therapy — Motivational Interviewing was developed to increase self-efficacy and motivation for drinking, and Cognitive Behavioral Therapy allows for individuals to develop strategies for drinking reduction. Both are evidence-based interventions that have been combined in previous studies for drinking reduction in problem drinkers.
  Other Names: MBSCT
  Arms: AD with physiological withdrawal (AD-W)
Drug: Naltrexone — Participants, who choose medication treatment, will be offered naltrexone (50 mg per day), which is an FDA-Approved medication for alcohol use disorder. According to the package insert for NTX, the medication has been associated with liver toxicity at very high doses (up to 300 mg/day); however, a number of clinical trials and published studies suggest there are few serious adverse effects, including minimal hepatotoxicity, associated with daily dose of 50 mg of naltrexone. Its most common side effects in opioid-free individuals are nausea, vomiting, anxiety, headache, abdominal discomfort, difficulty sleeping, fatigue, irritability, and decreased appetite. A rare serious adverse effect may include minimal liver toxicity, but is more likely to occur at very high doses (300 mg/day).
  Other Names: NTX
  Arms: AD with physiological withdrawal (AD-W); Problem Drinkers (PD)
Behavioral: Brief Advice — Brief Advice (BA) consists of a 20-minute session delivered by a study therapist, adhering to the NIAAA's Clinician Guide to Problem Drinkers. It includes personalized, normative feedback based on NIAAA drinking norms, goal selection, instructions on self-monitoring, discussion of drink reduction strategies, and distribution of the NIAAA bibliotherapy guide.
  Other Names: BA
Other: Referral to specialty substance use disorder treatment — Participants who present with complex drinking concerns will be referred to specialty substance use disorder treatment. This treatment will be provided in a separate treatment facility that focuses on substance use disorders and will potentially provide a combination of medication management and individual/group behavioral treatment for substance use disorders.
  Other Names: Referral
  Arms: AD with complex presentation (AD-CMPLX)

SUMMARY:
The purpose of this research study is to develop and test a care model to treat excessive drinking and alcohol use disorders in the primary care setting. The goal of this research study is to increase the identification and treatment of problem drinking in the primary care setting. Individuals will be asked to participate in this study because routine screening and assessment conducted at your primary care clinic indicates that you have recently exceeded healthy drinking limits as outlined by the National Institutes of Alcohol and Alcoholism.

DETAILED DESCRIPTION:
Excessive drinking (ED) and alcohol use disorders (AUD) remain one of the nation's leading public health problems, yet this problem is largely under-recognized and undertreated. Although many people with ED/AUD see a primary care physician annually, there has been limited research and implementation of models to treat ED/AUD in primary care. Important changes in the healthcare system and advances in alcohol research offer new and potentially transformative opportunities to integrate ED/AUD treatment into primary care practices. In particular, these changes have led to the development of new patient-centered, integrated care models that facilitate the treatment behavioral health issues in primary care. Experts have repeatedly called for the development of a chronic care model to treat alcohol problems in primary care, similar to models now used to treat other chronic illnesses, including depression. Yet, research to develop and test such models has been surprisingly limited. The primary aim of this study is to develop and test a chronic care model to treat ED/AUD in the patient-centered model home (PCMH) using the NIH stage model of intervention development. Specifically, using a mixed methods approach, this study proposes to adapt and test the collaborative care (CC) model for depression to treat ED/AUD in a high volume PCMH. Importantly, we will build the CC model onto a Screening, Brief Intervention, and Referral to Treatment (SBIRT) program that is already in place in the PCMH. Notably, this SBIRT model currently refers those with ED/AUD out to specialty treatment providers. The proposed study will be conducted in two phases. Phase I will involve initial adaptation of the CC model for depression. During this phase, relevant depression CC protocols and measures will be adapted for ED/AUD and piloted tested on participants (n = 25) recruited in a PCMH. Phase II will involve model refinement based on iterative cycles of patient and PCMH staff feedback and examination of drinking outcome data. During this phase, participants (n = 60) will be assessed and followed for three months. Iterative development will focus on: 1) utilizing a stepped-care model of treatment which will include outpatient detoxification, behavioral interventions, and medication intervention and management, 2) maximizing patient engagement, and 3) balancing the resource and expertise constraints of treating ED/AUD in a PCMH. Participants in Phases 1 and 2 will be followed at 1 and 3 months and primary outcome data on drinking outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Exceed NIAAA weekly or daily guidelines
* receive care at the 865 clinic
* are fluent in English
* are willing to provide signed, informed consent to participate
* available to complete research follow-ups
* are able to read English at the eighth grade or higher level and show no evidence of significant cognitive impairment

Exclusion Criteria:

* Meet DSM-V criteria for drug dependence other than for marijuana or nicotine
* on probation or parole
* have a serious psychiatric illness (e.g., psychotic disorder, bipolar disorder, severe major depression, etc.) that is likely to require pharmacologic treatment or that is currently treated with psychotropic medication; organic mood or mental disorders, or substantial suicide or violence risk

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Problem Drinkers (PD): PD will be offered a choice of either an evidence-based behavioral intervention(Motivational Enhancement Therapy) or medication (Naltrexone) plus medication management. These participants will also receive follow up assessments.
  Naltrexone: Participants, who choose medication treatment, will be offered naltrexone (50 mg per day), which is an FDA-Approved medication for alcohol use disorder. According to the package insert for NTX, the medication has been associated with liver toxicity at very high doses (up to 300 mg/day); however, a number of clinical trials and published studies suggest there are few serious adverse effects, including minimal hepatotoxicity, associated with daily dose of 50 mg of naltrexone. Its most common side effects in opioid-free individuals are nausea, vomiting, anxiety, headache, abdominal discomfort, difficulty sleeping, fatigue, irritability, and decreased appetite. A rare serious adverse effect may include minimal liver toxicity, but is more likely to occur at very high doses (300 mg/day).
  Brief Advice: Brief Advice (BA) consists of a 20-minute session delivered by a study therapist, adhering to the NIAAA's Clinician Guide to Problem Drinkers.
- AD With Physiological Withdrawal (AD-W): AD-W will referred to outpatient detoxification as part of standard care, unless medically contraindicated, and will be offered medication (naltrexone) plus medication management as or an evidence-based behavioral intervention (Modified Behavioral Self-Control Therapy [MBSCT]) adapted from our two prior protocols. These participants will also receive follow up assessments.
  Modified Behavioral Self-Control Therapy: Motivational Interviewing was developed to increase self-efficacy and motivation for drinking, and Cognitive Behavioral Therapy allows for individuals to develop strategies for drinking reduction. Both are evidence-based interventions that have been combined in previous studies for drinking reduction in problem drinkers.
  Naltrexone: Participants, who choose medication treatment, will be offered naltrexone (50 mg per day), which is an FDA-Approved medication for alcohol use disorder. According to the package insert for NTX, the medication has been associated with liver toxicity at very high doses (up to 300 mg/day); however, a number of clinical trials and published studies suggest there are few serious adverse effects, including minimal hepatotoxicity, associated with daily dose of 50 mg of naltrexone.
  Brief Advice: Brief Advice (BA) consists of a 20-minute session delivered by a study therapist, adhering to the NIAAA's Clinician Guide to Problem Drinkers.
Period: Overall Study
Arm/Group | At-Risk Drinkers (AR) | Problem Drinkers (PD) | AD With Physiological Withdrawal (AD-W) | AD With Complex Presentation (AD-CMPLX)
Started | 6 | 10 | 9 | 2
Completed | 6 | 9 | 8 | 2
Not Completed | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | At-Risk Drinkers (AR) | Problem Drinkers (PD) | AD With Physiological Withdrawal (AD-W) | AD With Complex Presentation (AD-CMPLX) | Total
Number analyzed (Participants) | 6 | 10 | 9 | 2 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 10 | 8 | 2 | 24
  >=65 years | 2 | 0 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 1 | 1 | 14
  Male | 2 | 2 | 8 | 1 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 1 | 1 | 4 | 0 | 6
  AmIndian/Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 0 | 3
  Native Hawaiian/other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 3 | 7 | 3 | 1 | 14
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 10 | 9 | 2 | 27

OUTCOME MEASURES:

1. Primary Outcome: Weekly Change in Drinking
Description: We used to the Timeline Followback Interview to collect the average weekly number of standard drinks of alcohol (about 9 grams) consumed at baseline (8 weeks prior to study enrollment) and during the 12-week treatment period. The minimum score is zero. There is no maximum score. Higher negative scores reflect a greater reduction in drinking and better outcomes.
Time Frame: Baseline (8 weeks prior to study enrollment) and the 12-week treatment period
Population: We examined the change in average number of standard drinks consumed weekly during the baseline (8 weeks prior to study enrollment) and the 12-week treatment period.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Problem Drinkers (PD): PD will be offered a choice of either an evidence-based behavioral intervention(Motivational Enhancement Therapy) or medication (Naltrexone) plus medication management. These participants will also receive follow up assessments.
  Motivation Enhancement Therapy: Motivation Enhancement Therapy (MET) similarly allows for goal choice in treatment, and has been shown to be effective in treating a broad spectrum of drinking problems in both abstinent and non-abstinent goal conditions. The unique goals of MET (enhancing intrinsic motivation for change and facilitating development of a self-generated change plan).
  Naltrexone: Participants, who choose medication treatment, will be offered naltrexone (50 mg per day), which is an FDA-Approved medication for alcohol use disorder.
  Brief Advice: Brief Advice (BA) consists of a 20-minute session delivered by a study therapist, adhering to the NIAAA's Clinician Guide to Problem Drinkers. It includes personalized, normative feedback based on NIAAA drinking norms, goal selection, instructions on self-monitoring, discussion of drink reduction strategies, and distribution of the NIAAA bibliotherapy guide.
- AD With Physiological Withdrawal (AD-W): AD-W will referred to outpatient detoxification as part of standard care, unless medically contraindicated, and will be offered medication (naltrexone) plus medication management as or an evidence-based behavioral intervention (Modified Behavioral Self-Control Therapy [MBSCT]) adapted from our two prior protocols. These participants will also receive follow up assessments.
  Modified Behavioral Self-Control Therapy: Motivational Interviewing was developed to increase self-efficacy and motivation for drinking, and Cognitive Behavioral Therapy allows for individuals to develop strategies for drinking reduction. Both are evidence-based interventions that have been combined in previous studies for drinking reduction in problem drinkers.
  Naltrexone: Participants, who choose medication treatment, will be offered naltrexone (50 mg per day), which is an FDA-Approved medication for alcohol use disorder.
  Brief Advice: Brief Advice (BA) consists of a 20-minute session delivered by a study therapist, adhering to the NIAAA's Clinician Guide to Problem Drinkers. It includes personalized, normative feedback based on NIAAA drinking norms, goal selection, instructions on self-monitoring, discussion of drink reduction strategies, and distribution of the NIAAA bibliotherapy guide.
Arm/Group | At-Risk Drinkers (AR) | Problem Drinkers (PD) | AD With Physiological Withdrawal (AD-W) | AD With Complex Presentation (AD-CMPLX)
Number analyzed (Participants) | 6 | 8 | 9 | 2
score on a scale | -11.4 (4.1) | -22.2 (8.0) | -39.6 (33.5) | -29.3 (9.9)

ADVERSE EVENTS:
Time Frame: The time frame for monitoring adverse events is 12 weeks or from baseline until the 12 week follow-up
Arm/Group | At-Risk Drinkers (AR) | Problem Drinkers (PD) | AD With Physiological Withdrawal (AD-W) | AD With Complex Presentation (AD-CMPLX)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/10 | 0/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/9 | 0/2
Other Adverse Events (participants affected / at risk) | 0/6 | 0/10 | 0/9 | 0/2

LIMITATIONS AND CAVEATS:
Recruitment limitations yielded a small sample. Although outcome data are reported they should be interpreted in the context of the small sample size. We also conducted a qualitative analysis (n=24) of participants' engagement in and acceptability of alcohol treatment in a patient centered medical home.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2018-03-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT02885311/Prot_SAP_000.pdf
  • Informed Consent Form: General (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT02885311/ICF_001.pdf
  • Informed Consent Form: General (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02885311/ICF_002.pdf
  • Informed Consent Form: General (2016-12-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02885311/ICF_003.pdf